CLINICAL TRIAL: NCT03095235
Title: Dietary Riboflavin (Vitamin B-2) and Cornea Cross-Linking
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: PI left the institution
Sponsor: University of Missouri-Columbia (Other)
Collaborators: University of South Florida (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2006390
Record Dates: First submitted 2016-10-13; First posted 2017-03-29 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Keratoconus; Cornea Ectasia
Keywords: keratoconus; cornea ectasia
MeSH Terms: conditions — Keratoconus | interventions — Riboflavin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment with riboflavin (Experimental): Patients will take 400 mg dietary riboflavin per day and go outside without sunglasses for 15 minutes per day to evaluate the effects of riboflavin B2 and natural UV light from sun exposure on cornea cross linking and stabilization of ectatic disease.
  Interventions: Dietary Supplement: Dietary riboflavin

INTERVENTIONS:
Dietary Supplement: Dietary riboflavin — Dietary riboflavin is vitamin B2. It has been shown to be safe in children in the treatment of migraines at doses of 400 mg per day. There are no known documented side effects
  Other Names: Vitamin B2

SUMMARY:
Corneal ectasia is characterized by irregularity and thinning of the cornea, causing the cornea to bulge forward and cause distorted vision and impaired visual acuity. Corneal ectasia is a complication after refractive (LASIK) surgery. It is also the primary problem in keratoconus, a gradually progressive inherited condition that typically is manifested in young adulthood, more commonly in women. Treatment approaches to stabilize the cornea's shape include rigid contact lenses, surgical implantation of stiff plastic intrastromal corneal ring segments, a collagen cross-linking procedure and, in severe cases, cornea transplantation. The collagen cross-linking procedure involves topical application of a concentrated riboflavin (vitamin B2) solution after the corneal epithelium is scraped, followed by ultraviolet (UV) light exposure. UV light stimulates riboflavin to form new bonds (cross links) between the cornea's connective tissue, giving the cornea additional strength to maintain its shape and prevent the need for transplantation. The cost of one treatment using this system is $2,500 to $3,500. A small prospective study including 7 patients with keratoconus was started on a trial of oral riboflavin and 15 minutes of natural sunlight exposure daily. These patients reported no adverse effects and preliminary results showed corneal stabilization and/or corneal flattening in all 7 patients It is hypothesized that dietary riboflavin and natural sunlight is as effective in corneal crosslinking as the currently FDA approved Avedro therapy. If the clinical study confirms the investigators' early observations of the benefits of this approach, coupled with animal studies that document corneal cross-linking, the investigators will have data to pursue funding for larger clinical and animal studies. This has the potential to save millions of dollars in health care costs and ease the burden of treatment in patients who require therapy to induce corneal cross-linking to stabilize the cornea's shape.

DETAILED DESCRIPTION:
Corneal ectasia as a complication from refractive (LASIK) surgery as well as keratoconus is a slowly progressive condition that results in high patient morbidity. Treatment options aim to stabilize the shape of the cornea using rigid contact lenses, surgical insertion of stiff plastic intrastromal rings, corneal cross linking, and ultimately corneal transplant in severe patients. The recently FDA approved "Dresden Protocol" involves painful cornea scraping followed by application of concentrated Riboflavin, followed by immediate collagen cross linking with UV light exposure which results in shortening and thickening of the collagen fibrils, and therefore a stronger, stiffer cornea. Avedro has demonstrated an average cornea flattening (K max reduction) of 1.4 diopters and 1.7diopters in two different studies. The current cost of Avedro therapy is between $2500 -$3500 per treatment. This is considered to be an accepted medical procedure at this time and therefore is beginning to be covered by several insurance companies.To spare the patient the severe pain involved in the current procedure, and to avoid the high cost (Avedro is not covered by any medical insurance), the investigator started 7 patients with keratoconus from 2011-2015 in his private practice in Seattle on a trial of oral riboflavin (100 mg or 400 mg daily) and 15 minutes of sunlight exposure daily. No adverse effects have ever been reported with high-dose dietary riboflavin supplements. The results of this preliminary trial are remarkable. During follow-up from 6 months to 5 years, all 7 patients have had corneal stabilization and/or corneal flattening. One patient experienced flattening of the cornea by 1.5 Diopters, comparable to the best results of the Avedro system. A limited animal study was recently completed and published in Switzerland by Dr. Farhad Hafezi , M.D., PhD which was published in the Journal of Cataract & Refractive Surgery that confirmed corneal cross-linking occurs in response to riboflavin and UV exposure from the sun and proven to successfully crosslink. Our current clinical study would expand the promising preliminary findings to a larger sample size. This has the potential to save millions of dollars in health care costs and ease the burden of treatment in patients who require therapy to induce corneal cross-linking to stabilize the cornea's shape.

To date eye specialists in Brazil, Texas and other locations are beginning to treat patients with our protocol and finding similar successful results using 400 to 800mg dietary riboflavin and 15 to 45 minutes of sunlight exposure for a period of 3 to 6 months with successful results.

ELIGIBILITY:
Inclusion Criteria:

* patients identified as having keratoconus or post refractive cornea ectasia with astigmatism of 1.5 Diopters or greater.

Exclusion Criteria:

* Known sensitivity to riboflavin, sunlight.
* patients on medications with side effects of increased sunlight sensitivity should discuss participation with their prescribing provider prior to participation

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2021-03-08 (Actual); Study Completion 2021-03-08 (Actual)

PRIMARY OUTCOMES:
Degree of corneal steepening | 6 months
  Keratometry measures the degree of astigmatism of the cornea to monitor the degree of cornea steepening

SECONDARY OUTCOMES:
Best corrected visual acuity | 6 months
  Measures the best vision the patient is able to see at that time

CONTACTS AND LOCATIONS:
Overall Officials: John S Jarstad, MD, Principal Investigator — University of South Florida - Department of Ophthalmology
Locations (1):
- University of South Florida Department of Ophthalmology, Tampa, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jarstad JS.Mega-dose DIetary Riboflavin in the Treatment of Keratoconus, Post-Refractive Cornea Ectasia and Migraine. Has its Time Arrived? Archives of Clinical Ophthalmology 2021:1(1):20
- [Background] Wu D, Lim DK, Lim BXH, Wong N, Hafezi F, Manotosh R, Lim CHL. Corneal Cross-Linking: The Evolution of Treatment for Corneal Diseases. Front Pharmacol. 2021 Jul 19;12:686630. doi: 10.3389/fphar.2021.686630. eCollection 2021. PMID 34349648
- [Result] Torres-Netto EA, Abdshahzadeh H, Lu NJ, Kling S, Abrishamchi R, Hillen M, Hafezi NL, Koppen C, Hafezi F. Corneal crosslinking with riboflavin using sunlight. J Cataract Refract Surg. 2023 Oct 1;49(10):1049-1055. doi: 10.1097/j.jcrs.0000000000001241. PMID 37343287